CLINICAL TRIAL: NCT02734446
Title: Randomized Controlled Clinical Trial to Evaluate the Efficacy of Supplementation With L. Reuteri + Vit. D3 in Asthmatic Children
Brief Title: To Evaluate the Efficacy of Supplementation With L. Reuteri + Vit. D3 in Asthmatic Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Prof. Michele Miraglia del Giudice, Prof., University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTN_D3
Record Dates: First submitted 2016-03-18; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Asthma
Keywords: Bronchial Inflammation; Asthma; Childhood Asthma Control Test (C-ACT); Asthma Exacerbations
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reuterin D3 drops (Active Comparator): Lactobacillus reuteri DSM 17938 (108 CFU) + Vitamin D3 (400 IU) 5 drops/day for 3 months (Reuterin D3 drops)
  Interventions: Drug: Reuterin D3 drops
- Placebo (Placebo Comparator): The patients will receive 5 drops/day of placebo for 3 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Reuterin D3 drops — 5 drops/day for 3 months
  Other Names: Lactobacillus reuteri DSM 17938 + Vit. D3
  Arms: Reuterin D3 drops
Other: Placebo — 5 drops/day for 3 months
  Arms: Placebo

SUMMARY:
The purpose of this project is to evaluate in a randomized clinical trial, double-blind, controlled, the effects of a dietary supplement containing Lactobacillus reuteri DSM 17938 and vitamin D3 in reducing bronchial inflammation and improve asthma control in patients in children with mild / moderate persistent asthma .

DETAILED DESCRIPTION:
To evaluate if the supplementation for three months with Lactobacillus reuteri DSM 17938 (108 CFU) + Vitamin D3 (400 IU) result in a reduction of the degree of allergic bronchial inflammation, measured with the Fractional exhaled nitric oxide (FeNO) and with a series of markers of bronchial inflammation (measured at 'beginning and at the end of the treatment on exhaled condensate): Interleukin 2(IL-2); Interleukin 4 (IL-4); Interleukin 10(IL-10); Interferon γ (IFN-γ).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 6 and 14 years old, of both sexes
* Diagnosis of mild / moderate persistent asthma (GINA step 2/3)
* Allergy mite (Dermatophagoides farinae and pteronyssinus + + + / + + + +)
* Levels of vitamin 25 (OH) D <30 ng / ml
* Signature of the informed consent of one parent or a legal representative

Exclusion Criteria:

* Cardiovascular disease or systemic
* anatomical abnormalities
* Other respiratory diseases
* Taking probiotics and / or prebiotics in the previous 2 weeks
* Taking vitamin D or systemic corticosteroids within 4 weeks
* Participation in other clinical trials

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Reduction of allergic bronchial inflammation | Up to 3 months
  Reduction of FeNO values
Reduction of allergic bronchial inflammation | Up to 3 months
  Reduction of a series of markers of bronchial inflammation: IL-2; IL-4; IL-10; IFN-γ.

SECONDARY OUTCOMES:
Improvement of asthma control by C-ACT | Up to 3 months
  Improvement in asthma control assessed by:
  C-ACT (Scores > 19)
Improvement of asthma control by reduction of bronchodilator | Up to 3 months
  Improvement in asthma control assessed by:
  Reduction use of bronchodilator
Improvement of asthma control by improvement of FEV-1 | Up to 3 months
  Improvement in asthma control assessed by:
  Improvement of Forced Expiratory Volume in 1 second (FEV-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Second University of Naples, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Miraglia Del Giudice M, Maiello N, Allegorico A, Iavarazzo L, Capasso M, Capristo C, Ciprandi G. Lactobacillus reuteri DSM 17938 plus vitamin D3 as ancillary treatment in allergic children with asthma. Ann Allergy Asthma Immunol. 2016 Dec;117(6):710-712. doi: 10.1016/j.anai.2016.09.004. Epub 2016 Oct 6. No abstract available. PMID 27720582